CLINICAL TRIAL: NCT01379001
Title: Assessment of Cholinergic and Cognitive Function Using Pharmacologic ASL-Perfusion MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Tamara Fong, Assistant Scientist/Assistant Professor of Neurology, Hebrew SeniorLife
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: K23AG031320 (NIH)
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Cholinergic Function
Keywords: cholinergic function; aging; pharmacologic MRI
MeSH Terms: interventions — Scopolamine; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Young (Experimental): Young healthy controls, aged 21-35
  Interventions: Drug: Scopolamine; Drug: Placebo
- Older (Experimental): Older healthy controls, aged 65-80
  Interventions: Drug: Scopolamine; Drug: Placebo; Drug: Donepezil

INTERVENTIONS:
Drug: Scopolamine — Scopolamine 0.4mg IM x 1 dose; adjustment in older group for weight (0.4mg/70kg)
Drug: Placebo — IM or PO placebo
Drug: Donepezil — donepezil 5mg PO x 1
  Other Names: Aricept
  Arms: Older

SUMMARY:
This research study will look at how medications affect the pattern of blood flow in the brain. This study will use a special type of MRI (magnetic resonance imaging) scan called perfusion MRI to make measurements of cerebral (brain) blood flow. The medications we will use in this study are scopolamine (commonly used to treat motion sickness), mecamylamine (used to treat high blood pressure), and donepezil (used to treat memory loss). Cognitive testing will also be obtained, and correlated with the blood flow patterns in the brain.

DETAILED DESCRIPTION:
Project Summary: This research project will investigate the value of combined pharmacologic manipulation and arterial spin-labeled perfusion MRI (pharmacologic ASL-pMRI) as an in vivo probe of cholinergic function. Methods to investigate cholinergic function in vivo are needed to better understand the role of acetylcholine in the physiology of the cerebral cortex, and in cognitive processes in health and in disease states. In this study, pharmacologic ASL-pMRI will be used to characterize the normal cerebral perfusion response to cholinergic manipulation in young healthy subjects. Cognitive measures will also be obtained and correlated with cerebral perfusion changes. Pharmacologic ASL-pMRI and cognitive testing will then be used to study how the cholinergic response is altered with normal aging and in delirium

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* Any neurological condition, such as brain tumor, history of stroke, seizure disorder, attention deficit disorder, normal pressure hydrocephalus, dementia, traumatic brain injury
* Any major medical conditions, such a cancer, diabetes, glaucoma, prostate disease, uncontrolled hypertension
* antihistamine use
* tricyclic antidepressant use
* presence of metal in body, including pacemaker, defibrillator, neurostimulator, metal implants, or foreign metal objects such as bullets or shrapnel.
* anxiety or panic disorder
* history of claustrophobia
* pregnancy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow | 3 hours
  cerebral blood flow will be measured 3 hours after drug administration using Arterial spin-labeled perfusion MRI

SECONDARY OUTCOMES:
cognitive performance | 4 hours
  participants will undergo cognitive testing following drug administration and MRI acquisition

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Fong, MD, Principal Investigator — Hebrew Rehabilitation Center